CLINICAL TRIAL: NCT05480436
Title: Immunogenicity and Safety of Inactivated COVID-19 Vaccine Coadministered With 23-valent Pneumococcal Polysaccharide Vaccine and Quadrivalent Influenza Vaccine in Hemodialysis Population: a Multicentre, Randomised, Controlled, Phase 4 Trial
Brief Title: Immunogenicity and Safety of BBIBP-Corv Coadministered With PPV23 and IIV4 in Hemodialysis Population
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Hunan Provincial Center for Disease Control and Prevention (Other); Sichuan Center for Disease Control and Prevention (Other Government); Guizhou Center for Disease Control and Prevention (Other); Xiangya Hospital of Central South University (Other); Beijing Institute of Biological Products Co Ltd. (Industry); Chengdu Institute of Biological Products Co.,Ltd. (Industry); Shanghai Institute Of Biological Products (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2022BBIBP-corv+IIV4+PPPV23
Record Dates: First submitted 2022-07-27; First posted 2022-07-29 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Hemolysis; COVID-19
MeSH Terms: conditions — Hemolysis; COVID-19 | interventions — COVID-19 Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental Group (Experimental): Total of 400 participants received one dose of BBIBP-Corv and IIV4 on Day 0, and received one dose of BBIBP-Corv and PPV23 on Day 28. Blood sampling was performed on Day 0, Day 28 and Day 56 for humoral immunity assessment.
  30 of the 400 participants were selected to collect three blood samples on Day 0, Day 42 and Day 56 for cellular immune assessment.
  Interventions: Biological: coadministration
- Control Group 1 (Active Comparator): Total of 400 participants received two doses of BBIBP-Corv on Day 0 and Day 28. Blood sampling was performed on Day 0, Day 28 and Day 56 for humoral immunity assessment.
  30 of the 400 participants were selected to collect three blood samples on Day 0, Day 42 and Day 56 for cellular immune assessment.
  Interventions: Biological: COVID-19 vaccine
- Control Group 2 (Active Comparator): Total of 400 participants received one dose IIV4 on Day 0 and received one dose PPV23 on Day 28. Blood sampling was performed on Day 0, Day 28 and Day 56 for humoral immunity assessment.
  Interventions: Biological: IIV4+PPV23

INTERVENTIONS:
Biological: coadministration — the coadministration of an inactivated COVID-19 vaccine (BBIBP-CorV) and IIV4 on Day 0, and the coadministration of BBIBP-CorV and PPV23 on Day 28
  Arms: Experimental Group
Biological: COVID-19 vaccine — received two doses of inactivated COVID-19 vaccine (BBIBP-CorV)
  Arms: Control Group 1
Biological: IIV4+PPV23 — received one dose of IIV4 on Day 0, and one dose of PPV23 on Day 28
  Arms: Control Group 2

SUMMARY:
Evaluation of immunogenicity and safety of inactivated COVID-19 vaccine (BBIBP-Corv) coadministered with PPV23 and IIV4 in hemodialysis population.

DETAILED DESCRIPTION:
Participants aged ≥18 undergoing hemodialysis were recruited and randomly assigned to one of three study groups.

Experimental Group : The participants received the first dose of BBIBP-Corv and IIV4 simultaneously on Day 0, and received the second dose of BBIBP-Corv and PPV23 simultaneously on Day 28.

Control Group 1: The participants received two doses of BBIBP-Corv on Day 0 and Day 28, respectively.

Control Group 2 : The participants received one doses of IIV4 on Day 0 and received one doses of PPV23 on Day 28.

Three blood samples were collected on days 0, 28 and 56 to test humoral immunity, and three blood samples were collected on days 0, 42 and 56 to test cellular immunity to SARS-CoV-2.

Any local or systemic adverse events after vaccination will be recorded.

ELIGIBILITY:
Inclusion Criteria 1 :

* Participants were hemodialysis patients aged ≥18 years.
* The duration of dialysis of the participants was ≥3 months.
* The life expectancy of participants was ≥2 years.
* Participants who have not previously been infected with SARS-CoV-2.
* Participants had not received any COVID-19 vaccine and had not received any influenza or pneumonia vaccine within 1 year.
* For female participants of reproductive age, they had no fertility plan within the first 3 months and had taken effective contraceptive measures within 2 weeks ; For male participants of reproductive age, no fertility plans were made within 3 months.
* Be able and willing to complete the entire study plan during the study follow-up period.
* Have the ability to understand the study procedures, voluntarily sign informed consent.

Inclusion Criteria 2 :

* Body temperature < 37.3 °C confirmed by clinical examination before enrollment .
* Systolic blood pressure (SBP) was < 160 mmHg and diastolic blood pressure (DBP) was< 100 mmHg , and fasting blood glucose (FPG) was ≤13.9 mmol/L on the day of enrollment.
* Female participants of reproductive age were not pregnant.

Exclusion Criteria 1 for the first dose:

* Being allergic to any component of vaccines and a history of severe allergic reactions to any vaccine or allergic to pollen, food and other common allergens, or a history of allergic reaction to eating eggs or using gentamicin sulfate.
* Participants with uncontrolled epilepsy or a history or family history of epilepsy, a history of Guillain-Barre syndrome, Reye syndrome, and other progressive diseases.
* Participants were confirmed to be infected with H1N1, H3N2, BY and BV influenza viruses within 6 months.
* Pregnant and lactating women.
* Participants were in the period of acute illness or acute onset of chronic disease, and the acute complication has been cured for less than two weeks.
* Participants with acute febrile diseases and infectious diseases (including hepatitis B, hepatitis C, HIV patients and carriers, as well as patients with suspected pulmonary tuberculosis symptoms such as hemoptysis, night sweats and weight loss).
* Participants with congenital immunodeficiency or currently receiving immunosuppressive therapy (oral steroid hormones, calcineurin inhibitors (CNIs), rituximab, long-term glucocorticoid use ≥1 week).
* Participants injected with non-specific immunoglobulin within 30 days.
* Participants received attenuated vaccines within 30 days and inactivated or other vaccines within 14 days.
* Serious drug adverse reactions and drug-related complications occurred during dialysis treatment.
* Participants with severe cardiovascular diseases (e.g., myocardial infarction, heart failure, malignant arrhythmia).
* Participants with infectious, suppurative and allergic skin diseases or severe skin itching (refers to the widespread and persistent attack; Affecting self-regulated activities of daily living or sleep; Systemic glucocorticoid or immunosuppressive therapy is required).
* Participants with malignant tumors.
* Participants had a history of seizures, encephalopathy, or psychiatric disorders (depressive mania, depression, schizophrenia, etc.).
* Other Participants whose physical conditions, as determined by the investigator, are not suitable for inclusion in clinical studies.

Exclusion Criteria 2 for the first dose:

* Participants who need medical intervention (except blood glucose) after laboratory tests (blood routine, blood biochemical, coagulation routine) are judged by the investigator.
* Participants had a history of clearly diagnosed thrombocytopenia or other coagulation disorders, which may be contraindicated as subcutaneous injections
* The participant did not inform the investigator in time of any condition mentioned in " Exclusion Criteria 1 for the first dose ".
* Other Participants whose physical conditions, as determined by the investigator, are not suitable for inclusion in clinical studies.

Exclusion criteria for the second dose:

* Subjects who had vaccine-related serious adverse reactions after vaccination.
* High fever (axillary temperature > 40.0℃) lasted for two days after vaccination, or severe allergic reaction occurred.
* Any vaccine-related neurological adverse reactions occurred after vaccination.
* Participants experienced new conditions that met the "exclusion criteria for the first dose ".
* Other reasons for exclusion considered by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2022-08-05 (Actual); Primary Completion 2023-01-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Seroconversion rate against SARS-CoV-2 | 28 days after two doses vaccination (Day 56)
  The rate of seroconversion against SARS-CoV-2
Seroconversion rate against IIV4 | 28 days after vaccination (Day 28)
  The rate of seroconversion against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
Seroconversion rate against PPV23 | 28 days after vaccination (Day 56)
  The rate of seroconversion against 23 pneumococcal serotypes
Neutralizing antibody GMT against SARS-CoV-2 | 28 days after two doses vaccination (Day 56)
  Neutralizing antibody GMT against SARS-CoV-2 after vaccination
Hemmagglution inhibition antibody GMT against IIV4 | 28 days after vaccination (Day 28)
  Hemmagglution inhibition antibody GMT against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
IgG antibody GMC against PPV23 | 28 days after vaccination (Day 56)
  IgG antibody GMC against 23 pneumococcal serotypes
Neutralizing antibody geometric mean increase (GMI) against SARS-CoV-2 | 28 days after two doses vaccination (Day 56)
  Neutralizing antibody GMI against SARS-CoV-2 after vaccination
Hemmagglution inhibition antibody GMI against IIV4 | 28 days after vaccination (Day 28)
  Hemmagglution inhibition antibody GMI against influenza A (H3N2, H1N1) type and B (BY, BV) type viruses
IgG antibody GMI against PPV23 | 28 days after vaccination (Day 56)
  IgG antibody GMI against 23 pneumococcal serotypes

SECONDARY OUTCOMES:
Adverse events rate | 0-7 days or 0-28 days following vaccinations
  Analyse the incidence of adverse events following vaccination, both solicited and unsolicited
Serious adverse event rate | 0-6 months
  Report and analyse serious adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Tao Huang, Principal Investigator — Hunan Provincial Center for Disease Control and Prevention
Locations (3):
- China (3):
  - Xiangya Hospital Central South University, Changsha
  - Sichuan Center for Disease Control and Prevention, Chengdu
  - Guizhou Center for Disease Control and Prevention, Guiyang

IPD SHARING:
Plan to Share IPD: No